CLINICAL TRIAL: NCT04776538
Title: A Single-centre, Double-blinded, Randomised, Placebo-controlled, Phase II Study to Investigate the Safety and Efficacy of Mesenchymal Stem Cell for Radiation-induced Hyposalivation and Xerostomia in Previous Head and Neck Cancer Patients (MESRIX-III)
Brief Title: Safety and Efficacy of Mesenchymal Stem Cell for Radiation-induced Hyposalivation and Xerostomia in Previous Head and Neck Cancer Patients
Acronym: MESRIX-III
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Cardiology Stem Cell Centre, The Heart Centre, Rigshospitalet (Unknown); Department of Oncology Herlev Hospital, Denmark (Unknown); Department of Dentistry and Oral Health, Aarhus, Denmark (Unknown)
Responsible Party: Principal Investigator, Kathrine Kronberg Jakobsen, Medical Doctor, investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVB2018-1
Record Dates: First submitted 2021-01-21; First posted 2021-03-01 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Xerostomia Following Radiotherapy
Keywords: stem cell; Adipose derived stem cell

STUDY DESIGN:
Intervention Model Description: The study is a prospective, double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: The sponsor, investigators, study staff (except for staff involved in stem cells preparation and staff involved in bioanalytical analyses) and patients will be blinded to treatment assignment and care will be taken to ensure the study team is kept blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell group (Experimental): 60 patients will be randomized to receive adipose-derived allogeneic stem cells
  Interventions: Biological: Stem cells
- Placebo group (Placebo Comparator): 60 patients will receive placebo consisting of CryoStor10 (BiolifeSolutions), the freeze media for ASCs containing 10% Dimethyl sulfoxide (DMSO).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Stem cells — Each participant will be double-blindly randomized to receive either adipose-derived allogeneic stem cells or placebo consisting of CryoStor10 (BiolifeSolutions), the freeze media for ASCs containing 10% Dimethyl sulfoxide (DMSO).
  Arms: Stem cell group
Biological: Placebo — Each participant will be double-blindly randomized to receive either adipose-derived allogeneic stem cells or placebo consisting of CryoStor10 (BiolifeSolutions), the freeze media for ASCs containing 10% Dimethyl sulfoxide (DMSO).
  Arms: Placebo group

SUMMARY:
The incidence of head and neck cancer is increasing in the Western World, including Denmark. Cancer of the head and neck and its treatment often have a detrimental and lifelong impact on the quality of life of the patients. Radiotherapy is a key component for approximately 80% of all patients with head and neck cancer and despite the enormous improvement in ionizing radiotherapy, the radiation still leads to significant ionizing of healthy tissue, including the radiation-sensitive salivary glands. Salivary glands suffer severe damage from radiation, and as these cells are the principal sites of fluid secretion one of the most prevalent side effect of irradiation for head and neck cancer is hyposalivation and dry mouth syndrome, xerostomia. Xerostomia leads to debilitating oral disorders and major implication for the overall quality of life, including social life and professional life. Currently, only symptomatic treatment is available to patients suffering from xerostomia, and therefore there is an immense, unmet need for new treatment strategies for hyposalivation and xerostomia.

Stem cells have been identified as a potential treatment modality for a wide variety of disorders by their ability to differentiate into many functional cell types, and stem cells have been suggested as an approach to restoring the function of salivary glands after radiotherapy damage.

The purpose of the study is to assess the efficacy and safety of the injection of stem cells from healthy donors on radiation-induced salivary gland hypofunction and xerostomia in previous head and neck cancer patients. The project can potentially help to develop a clinically relevant treatment option for the growing number of patients suffering from xerostomia after irradiation. The development of new therapies is especially meaningful since only sub-optimal, symptomatic treatments are currently available, and since the symptom of xerostomia immensely reduces quality of life.

DETAILED DESCRIPTION:
Background:

Xerostomia is the diagnosis of the subjective feeling of dry mouth. Xerostomia can coexist with or exist without a reduced production of saliva, although xerostomia is first perceived when unstimulated whole saliva flow rate is reduced by more than 40-50%. In this context, a subnormal or pathologically reduced saliva production (hyposalivation) will severely diminish the quality of life and lead to severe dental decay. The two main causes of grave xerostomia are Sjögren's syndrome and radiation therapy for head and neck cancer. Radiation therapy plays a central role in the curative treatment of most upper head and neck cancers, either as a single modality or in combination with chemotherapy and/or surgery, and the prevalence of xerostomia after head and neck radiation ranges from 74 to 85%.

Radiation therapy increases local tumor control significantly along with the chance of survival, but despite the more advanced methods of radiation therapy, Intensity-Modulated radiation therapy (IMRT), a significant proportion of the radiation is deposited in the healthy tissue surrounding the tumor. The decrease of saliva secretion after radiation therapy predisposes the patients to a variety of conditions. These are either directly or indirectly a result of the decreased production of saliva and include xerostomia, impairment of the normal oral functions (talking, chewing, and swallowing) due to insufficient wetting, and reduced lubrication of mucosal surfaces and the ingested food which impairs nutrition. Furthermore, the oral mucosa can become dry, making the oral mucosa vulnerable, which may lead to frictional trauma and ulceration. In addition, a reduced salivary flow results in a reduced "rinsing" of the entire oral cavity, thus leading to microbial overgrowth, which in addition to other factors may result in rapid dental decay, dental erosion, and oral candidiasis (thrush).

Stem cells have been identified as a potential treatment modality for a wide variety of disorders by their ability to differentiate into many functional cell types. For more than ten years, researchers have investigated the potential of mesenchymal stem cells (MSCs) as an approach to restoring the function of salivary glands after radiotherapy damage and several groups have addressed the use of MSCs or adipose-derived mesenchymal stem cells (ASCs) in preclinical studies of radiation-induced salivary gland dysfunction.

The research group has completed an encouraging randomized-controlled pilot study (MESRIX-I) with 30 patients assessing the safety and efficacy of ex-vivo expanded autologous ASCs for radiation-induced xerostomia in an effort to regenerate the function of the salivary glands (EudraCT nb:2014-004349-29). The results of this study show most importantly that the treatment is safe without any serious adverse events (SAE) and no systemic reactions, and secondly, the patients treated with stem cells have a promising enhanced production of saliva of 33%-50%. Furthermore, the research group has shown that the stem cell group gained vital quality of life measures compared with the placebo group in the form of diminished trouble in eating.

The research group has furthermore recently investigated the safety of allogenic ASCs for the treatment of xerostomia (MESRIX-II) with a clinical safety and feasible trial (EudraCT nb: 2018-003856-19). The study included ten patients who received intraglandular injections of allogeneic ASCs. No serious treatment-related adverse reaction occurred, and the efficacy data was similar to the results from our first trial with autologous ASCs.

Research hypothesis Treatment with ASCs will result in an improvement of the participant's unstimulated and stimulated whole saliva flow rate and ameliorate the xerostomia and increase quality of life.

Study aim The purpose of the study is to assess the efficacy and safety of the injection of allogeneic ASCs from healthy donors on radiation-induced salivary gland hypofunction and xerostomia in previous head and neck cancer patients. The project can potentially help to develop a clinically relevant treatment option for the growing number of patients suffering from xerostomia after irradiation. The development of new therapies is especially meaningful since only sub-optimal, symptomatic treatments are currently available, and since the symptom of xerostomia immensely reduces quality of life.

Study design The study is an investigator-initiated, prospective, single-center, double-blinded, randomized, placebo-controlled trial to compare the safety, tolerability and efficacy of ASCs as a treatment for radiation-induced hyposalivation and xerostomia for previous head and neck cancer patients.

Method Patients between the age of 18-70 years previously treated with radiation for a head and neck cancer and a clinically evaluated reduced salivation and hyposalivation, evaluated by a screening, can be included. Each participant will be double-blindly randomized to receive either allogeneic ASCs or placebo consisting of CryoStor10 (BiolifeSolutions), the freeze media for ASCs containing 10% Dimethyl sulfoxide (DMSO). Allogeneic ASCs are provided from the Cardiology Stem Cell Centre (CSCC) at Rigshospitalet.

Patients will be evaluated on salivary gland function and saliva flow rate by sialometry. Both unstimulated whole saliva and stimulated whole saliva will be collected. Furthermore, the investigators will analyze the following on the collected saliva: pH and bicarbonate by ionic balance estimation, sodium, potassium, calcium, phosphate, chloride and fluoride, total protein and selected proteins, and amylase. For evaluation of the participants´ perception of xerostomia, the participants will answer validated questionnaires in Danish (EORTC QLQ Module for H&N-35 and XQ) at baseline and after four months. These patient-reported outcomes (PRO) questionnaires are essential, validated tools for estimating the degree of quality of life (QoL) and xerostomia.

Recruitment of MESRIX-III participants and obtaining informed consent MESRIX-III participants (recipients/placebo) will be recruited through the Department of Otolaryngology, Head and Neck Surgery at Rigshospitalet and Oncology Departments at Rigshospitalet and Herlev Hospital, and through our databases on head and neck cancer patients. The investigator will send a letter to eligible patients who have been treated and followed for their previous cancer disease. Eligible patients can also contact the investigators or a trained member of the MESRIX-III study by phone or by a specific study e-mail (regionh-stamcelle.rigshospitalet@regionh.dk) if the eligible patients wish to receive a letter with further information. Subsequently, the principal investigator or a trained member of the MESRIX-III study group will contact patients by phone and inquire about their interest in participating in the research project.

If the eligible patients have an interest in participating in the project, the eligible patients will be invited to an interview at the outpatient clinic of the Department of Otolaryngology, Head and Neck Surgery, Rigshospitalet for further information concerning the trial. In the written information material, besides material about the trial, the pamphlets "Rights of test subjects in a health scientific research project" and "before decision" will be included. The right to bring counsel to the information interview will likewise be explained. Motivated patients referred from doctors in other parts of Denmark and patients who approach our department with an interest in participation in the stem cell research will also be offered information about the trial. Patients from all parts of Denmark can be included if the participants pass the inclusion and exclusion criteria described below. However, transportation and accommodation cannot be provided.

The information interview will take place in an undisturbed environment with the principal investigator or trained member of the MESRIX-III study group, who has the professional qualifications to communicate the content of the research project, and who will clearly explain that it is a request to participate in a health science research project. The participant will be given oral information about the project in layman's terms on the basis of the written information, and any questions will be answered. The oral information will be adapted to the participant's requirements, and it will be explained without the use of technical terms. Participants will be informed of the right to reflection following the information interview. Participants will likewise be informed of the opportunity to get feedback on the scientific results but will also be informed that no new information on the individual participant's disease or prognosis will be obtained. The potential participants for MESRIX-III will be contacted by telephone by the responsible physician for final commitment to participate. If participants are still interested in participating in the project, an appointment is made where a medical history is taken, and where the remaining trial appointments will be planned in agreement with the participant, and here the participants and the responsible physician will sign the medical consent form.

Evaluation, reporting, and recording of adverse events All adverse events (AEs) are monitored and recorded along with concomitant medicine at the scheduled follow-up (day one, and 4 months after the intervention). AEs are defined as any untoward medical occurrence in the clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with the treatment (ASC/placebo). AEs will be assessed and graded according to Common Terminology Criteria for Adverse Events v5.0 guidelines (CTCAEv5.0). Thus, all adverse events are recorded with CTCAE grade. All grade 3 and grade 4 events and incidents considered related to this trial will be reported to the sponsor by the investigator immediately after the events are discovered.

An adverse reaction (AR) is defined as any untoward or unintended response in a participant to an investigational medical product (IMP) which is related to any dose administered to that subject.

An adverse Drug Reaction (ADR) is stated as all noxious and unintended responses to a medicinal product related to any dose should be considered ADR.

Serious Adverse Event (SAE), Serious Adverse Reaction (SAR), or Suspected Unexpected Serious Adverse Reaction (SUSAR), means any AE, AE, SUSAR, respectively, that:

1. Results in death or
2. A serious deterioration in health that

   1. Resulted in life-threatening illness or injury
   2. Required hospitalization or prolongation of existing hospitalization
   3. Resulted in permanent impairment of body structure or body function
   4. Resulted in medical or surgical treatment to prevent the above
3. Lead to foetal death, congenital anomaly or birth defect, or other negative effect on the foetus
4. Anything the Principal Investigator deems to be of Clinical serious significance

Medical judgment will be exercised by the primary investigator together with the sponsor whether an AE or AR should be classified as serious in other situations.

The included participants will be instructed to contact the principal investigator or a special trained person from the research group in case of events with possible relation to the trial treatment within the main study period.

The principal investigator will immediately (within maximum 24 hours after receiving the information) inform the sponsor if SAR, SAE or serious suspected adverse reactions occurs. The sponsor will report SUSAR (Suspected Unexpected Serious Adverse Reaction) to the Danish Medicines Agency and the Danish National Committee on Health Research Ethics within 15 days of occurrence and 7 days in case of death or life-threatening issue. Unexpected reactions are defined as reactions that are not described in the section "Reference Safety information" of this protocol. All other unexpected serious adverse reactions will be reported within 15 days after the sponsor becomes aware of these.

All SARs that have occurred during the trial will be reported to The Danish Medicines Agency, The Danish Patient Safety Authority, and the National Committee on Health Research Ethics (if appropriate) once a year by the sponsor.

The sponsor will annually send a concise review and evaluation of pertinent safety information, a Development Safety update report (DSUR) collected during the reporting period related to the Danish Medicines Agency (DKMA).

After completion of the trial, the sponsor will after 90 days inform the Danish Medicines Agency that the study is completed. Within a year, the sponsor will submit trial results to the board, according to the law on drugs (Lov om lægemidler) § 89. 2, No. 4

Reference safety information (RSI) Adverse events with possible relation to injection of ASCs: Type; Frequency; Seriousness Temporary soreness of the salivary gland; 10-50%; Not serious Temporary redness of the salivary gland; 10-50%; Not serious Temporary swelling of the salivary gland; 10-50%; Not serious

Adverse events with relation to similar procedures and in MESRIX-I: Type; Frequency; Seriousness Temporary soreness of the salivary gland (up to 7 days after injection); 10-20%; Not serious Temporary redness of the salivary gland (up to 7 days after injection); 10-20%; Not serious Temporary swelling of the salivary gland (up to 7 days after injection); 10-20%; Not serious Infection of the salivary gland; 0.5-5%; Not serious Bleeding/hematoma in the salivary gland; 1-5%; Not serious

The above numbers and AEs are based on the previous phase I-II trial (EudraCT: 2014-004349-29) and on the literature cited and described in the section "Risk Assessment". In the previous study by the research group, MESRIX-I, with autologous ASCs no SAR or SUSARs were detected, so any SAR in this study will be reported as a SUSAR.

Long-term safety and efficacy follow-up Following Committee for Medicinal Products for Human Use (CHMP) under EMEA draft from January 2018 on safety and efficacy (S&E) follow-up and risk management of advanced therapy medicinal products (ATMP), the MESRIX-III participants will be invited to a follow-up of efficacy and ARs one year after the intervention (ASCs/placebo). Longer follow-up is not needed based on the reported long-term safety described in the section.

"Risk Assessment". Follow-up will include basic ear, nose, and throat examination, fiberscope, ultrasound of submandibular glands, sialometry, and blood samples. Data from the electronic medical journals and national pathology database will be gathered. It is expected that a number of the participants will have a recurrence of their primary cancer during the study or follow-up period due to the nature of the head and neck cancer. The allogeneic MSCs are believed to be rejected in the recipients, and the stem cells are adult non-pluripotent. However, in case of recurrence of cancer or new primary cancer developments each case will be carefully evaluated and potentially investigated with genetic analysis in an attempt to distinguish whether a tumor is due to recurrence, the administered product, or endogenous tumor formation.

Sample size and power considerations From MESRIX-I it appeared to be realistic to increase saliva production for whole unstimulated salivary flow (in milliliter(ml)/minut) rate by about 33% or in absolute numbers from 0.125 to 0.151 after 1 month and 0.155 after 4 months. The power calculation is based on a power of 0.8 and an alpha of 0.05. This means that the total number of patients included would have to be 100 (50 in each group) for a paired t-test. 10-20 additional participants may be included to compensate for dropout during the study period. The investigators believe that a 33% increase in whole, unstimulated salivary flow rate is clinically important and also realistic to detect.

Ethical considerations The trial is conducted in accordance with the Helsinki II declaration. The National Committee on Health Research Ethics and the Danish Data Protection Agency (DPA) will be requested permission to conduct the study. Moreover, the Danish Medicines Agency will be requested approval, and the trial will be monitored by the Good Clinical Practice (GCP) unit (Birgitte Grøn). Each volunteer (MESRIX-III participants) is required to give written informed consent before he/she can be included in the study. Information obtained about participants' health, other purely private matters, and other confidential information is covered by professional secrecy. No project participant has a personal financial incentive to implement the described project. The samples will be analyzed and stored in Denmark.

Risk assessment When the study participants in MESRIX-III will receive either ASCs or placebo into the large salivary glands the risk of adverse events such as infection and bleeding is estimated to be below 0.5% when using similar procedures. In our previous studies, none of the 40 participants developed adverse reactions.

The MESRIX-III participants may also experience some pain briefly during injection of the transplant product (ASCs or placebo).

A theoretical risk of a possible carcinogenic effect in the treatment of MSC/ASCs has been discussed. This is due to their production of growth factors such as epidermal growth factor (EGF), a factor produced by the MSC/ASCs. These considerations are particularly relevant since ASCs are used in participants previously diagnosed with cancer. However, in model systems of cancer, the effect of MSCs on cancer growth is controversial as MSCs have both been shown to be inhibitory and stimulatory. Further, numerous clinical trials with more than 1000 participants have been conducted with MSCs in different participant populations, and no increase in the incidence of cancer has been detected. These studies include local injection of MSCs. With respect to the use of ex vivo expanded MSCs, despite extensive research, there is no data indicating malignant transformation of expanded human MSCs/ASCs.

Data collection Source data: There will be source documentation for all data in Case Report Form (CRF).

The study director allows direct access to study data and study documents for the monitoring, audit, and inspection of the Science Ethics Committee, the Danish Health and Medicines Authority, or similar authorities in other countries. Permission will be sought from the DPA for the processing of personal data under the General Data Protection Regulation. Applications will be sent via the legal secretariat, Rigshospitalet.

Data will be analyzed with R. Our data will be kept securely in the electronic data capture system (EDC) Redcap. All data will be directly entered. The trial will be completed when all data is collected.

All results will be stored and analyzed electronically; participants' anonymity is ensured in accordance with the national data legislation. After completion of the study, data will be stored in an anonymous form. Data containing social security numbers will be kept locked and inaccessible to unauthorized persons.

Subject confidentially The investigator is obliged to ensure that participant anonymity is protected and maintained. On the CRF´s subjects should be identified by their initials and a subject study number only, Documents that are not for submission (e.g., signed informed consent forms) will be kept in strict confidence by the principal investigator. In compliance with the GCP Guidelines, it is required that the investigator and the institution permit authorized representatives of a monitoring company direct access to reviewing subjects' original medical records for verification of study-related procedures and data. All information obtained concerning this protocol regarding participants is protected according to the General Data Protection Regulation (GDPR).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years
2. Previous radiotherapy +/- chemotherapy for head and neck cancer 2 years' follow-up without recurrence
3. Clinically reduced salivation and hyposalivation, evaluated by a screening
4. Unstimulated salivary flow rate between 0.2 milliliter(mL)/minut (min) and 0.05 mL/min
5. Grade 1-3 xerostomia as evaluated by the UKU side effect rating scale
6. World Health organization (WHO) Performance status (PS) 0-1 59
7. Informed consent

Exclusion Criteria:

1. Any cancer in the previous 4 years (not including the head and neck cancer and basocellular carcinomas)
2. Xerogenic medications
3. Penicillin or Streptomycin allergy
4. Any other diseases of the salivary glands, e.g. Sjögren's syndrome or sialolithiasis
5. Previous submandibular gland surgery
6. Previous treatment with any type of stem cells in the saliva glands
7. Pregnancy or planned pregnancy within the four months study period
8. Breastfeeding
9. Smoking within the previous 6 months.
10. Alcohol abuse (consumption must not exceed 7 units/week for women and 14 units/week for men (Danish National board health alcohol guidelines)
11. Any other disease/condition judged by the investigator to be grounds for exclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Salivary gland function | 4 month
  Change in salivary gland function measured by a 4 months change in unstimulated whole saliva flow rate in the group receiving ASCs compared with the group of participants receiving placebo (control group receiving injections of CryoStor10 (BiolifeSolutions), the freeze media for ASCs).

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 4 month
  Safety evaluated by the incidence of adverse events at four months.
Patient-Reported Outcome of xerostomia | 4 month
  For evaluation of the participants´ perception of xerostomia, the participants will answer validated questionnaires in Danish at baseline and after four months. Patients will fill out EORTC QLQ Module for H&N-35 (evaluates overall implications of the xerostomia)
Patient-Reported Outcome of xerostomia | 4 month
  For evaluation of the participants´ perception of xerostomia, the participants will answer validated questionnaires in Danish at baseline and after four months. Patients will fill out the Xerostomia Questionnaire (XQ: self reported symptoms)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring pH.
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring bicarbonate level by ionic balance estimation
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of sodium (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of potassium (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of calcium (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of phosphate (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of chloride (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of fluoride (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of total protein (mmol/L)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of fluoride (ppm)
Salivary composition | 4 month
  Change in the composition of saliva after four months by measuring level of amylase (U/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Christian von Buchwald, MD, DMSc, Professor, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlander AF, Jakobsen KK, Jersie-Christensen R, Hansen J, Bendtsen SK, Kastrup J, Belstrom D, Lynggard CD, Gronhoj C, von Buchwald C. Exploring the salivary proteome following intraglandular mesenchymal stromal cell therapy for radiation-induced hyposalivation in previous head and neck cancer patients: a secondary study protocol for the MESRIX-III, randomised, controlled trial. Trials. 2025 Nov 28;26(1):554. doi: 10.1186/s13063-025-09074-4. PMID 41316394
- [Derived] Jakobsen KK, Carlander AF, Gronhoj C, Todsen T, Melchiors J, Paaske N, Madsen AKO, Kastrup J, Ekblond A, Haack-Sorensen M, Farhadi M, Maare C, Friborg J, Lynggard CD, von Buchwald C. Effectiveness and safety of mesenchymal stem/stromal cell for radiation-induced hyposalivation and xerostomia in previous head and neck cancer patients (MESRIX-III): a study protocol for a single-centre, double-blinded, randomised, placebo-controlled, phase II study. Trials. 2023 Sep 1;24(1):567. doi: 10.1186/s13063-023-07594-5. PMID 37658468